CLINICAL TRIAL: NCT03171636
Title: Analysis of the Types and Frequency of EGFR and KRAS Mutations and Clinical-prognostic Correlation in Brazilian Lung Cancer Patients at Erasto Gaertner Hospital, Curitiba, Brazil.
Brief Title: Frequency of EGFR and KRAS Mutations and Clinical-prognostic Correlation in Brazilian Lung Cancer Patients
Status: Completed | Type: Observational
Sponsor: Hospital Erasto Gaertner (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Thais Abreu de Almeira, MD, Hospital Erasto Gaertner
Other Study IDs: HEG02
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Lung Neoplasms; KRAS Gene Mutation; EGFR Gene Mutation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA sample from formalin-fixed paraffin-embedded (FFPE) tissue.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The assessment of the type and frequency of EGFR and KRAS mutations in lung cancer patients, as well as clinical-prognostic correlation, are crucial in the era of targeted therapies. EGFR-activating mutations predict responsiveness to EGFR tyrosine kinase inhibitors (TKIs) in non-small cell lung cancer (NSCLC) patients and KRAS analysis will be useful in a near future for newest target drugs. In Brazil, few data about the prevalence of EGFR and KRAS mutations is available and their knowledge would allow optimize personalized medicine.

DETAILED DESCRIPTION:
Assessment of the types and frequency of EGFR and KRAS mutations in NSCLC, as well clinical-prognostic correlations has been extensively studied in many populations. Few Brazilian studies evaluating mutational status in NSCLC has been done so far, none of then explored the regional background nor have considered the quantitative analysis of mutant cell in each sample. Quantitative analysis of the tumor maybe relevant for treatment design for positive samples, p.e a tumor with 90% of mutant clones versus a 15% of mutant clones, which can be obtained currently by the method of pyrosequencing. In this study, investigators will assess EGFR and KRAS status through the pyrosequencing quantitative technique, and will also correlate these with clinical-pathological variables among both adenocarcinoma and squamous cell histological subtypes. So far, no study that have made this correlation is available.

ELIGIBILITY:
Inclusion Criteria:

* Brazilian patients with metastatic non-small cell lung cancer.

Exclusion Criteria:

* Small cell lung cancer and non-metastatic patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From 237 patients with NSCLC treated at Erasto Gaertner Cancer Hospital, the largest reference cancer hospital in the Southern Brazil, from January 2005 to January 2017, we could select 130 FFPE specimens stored at the Pathology Department.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
EGRF mutation status | 3 years
  results of presence or absence in all tumor samples (FFPE) obtained from patients
KRAS mutation status | 3 years
  results of presence or absence in all tumor samples (FFPE) obtained from patients

CONTACTS AND LOCATIONS:
Overall Officials: Thais A Almeida, MD, Principal Investigator — Liga Paranaense de Combate ao Cancer
Locations (1):
- Hospital Erasto Gaertner, Curitiba, Paraná, Brazil